CLINICAL TRIAL: NCT04362605
Title: Case Series of Combined Endoscopic Negative Pressure Therapy and Surgical Treatment of Anastomotic Insufficiencies After Oncological Gastrectomies
Brief Title: Endoscopic Negative Pressure Therapy After Oncological Gastrectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTuebingen
Record Dates: First submitted 2020-02-25; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-02

CONDITIONS: Anastomotic Leak Esophagus
Keywords: endoscopic negative pressure therapy

STUDY DESIGN:
Intervention Model Description: Patients after gastrectomy who suffer from anastomotic leak
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervenional group (Experimental): ENPT
  Interventions: Procedure: Endoscopic Negative Pressure Therapy

INTERVENTIONS:
Procedure: Endoscopic Negative Pressure Therapy — In patients with suspected insufficiency of the esophagojejunostomy first an index endoscopy under general anesthesia with endotracheal intubation was indicated. Standard gastroscopes with outer diameter of 9.8mm were used with carbon dioxide insufflation.
  Definition of a anastomotic leak were endoscopic or radiological dehiscences at the esophagojejunostomy with extravasation of fluids and gas. In cases of insufficiencies start of endoluminal ENPT were indicated.
  Decision criteria for placement of OPD or OFD were the defect size, radiological findings and clinical situation of the patient. A CT scan in patients with suspected EJAL was done in all cases.
  For endoluminal ENPT, the open-pore drainage system is placed within the lumen of the digestive tract at the entrance to the cavity.
  Other Names: Endoscopic Vacuum Therapy; Endoscopic Vacuum Assisted Closure

SUMMARY:
Background and study aims: Management of esophago-jejunal anastomotic leackages (EJAL) after gastric resections is challenging. Endoscopic negative pressure therapy (ENPT) is an emerging effective tool for treatment of gastrointestinal and anastomotic leaks. We use ENPT for EJAL after oncological gastric resections as first line therapy since 2018. The aim of the study was to present our results with this strategy by a case series.

Patients and methods: Eight patients were treated with ENPT for EJAL after oncological gastric resections between 01.2018 and 12.2019. A retrospective analysis of patient's and therapy related data was performed.

Results: Time of detection was 6.25 ± 2.54 days after surgery. After 15.63 ± 9.92 days of ENPT, 6.43 ± 3.66 endoscopies and 38.75 ± 17.35 days of hospitalization, endoscopic treatment with ENPT combined with minimal-surgery for sepsis-control was effective in seven of eight patients. In one patients treatment was changed to Stent-based therapy combined with further surgical interventions.

Conclusions: ENPT is one step in the complication management of patients with anastomotic insufficiencies after oncological gastric resections. It can be recommended in combination with minimal invasive surgery for sepsis-control. Success of ENPT for EJAL seams to be dependent on the age and size of the insufficiency and the clinical situation of the patient.

DETAILED DESCRIPTION:
Endoscopic negative pressure therapy (ENPT):

OPD: The commercially available Eso-SPONGE® System (B. Braun Melsungen AG, Melsungen, Germany) was used for endoluminal vacuum therapy. For positioning the OPD in loop-technique a loop (MersileneTM, Polyester, 4 Ph. Eur., Ethicon®, Norderstedt, Germany) is fixed at the distal end of the drainage, gripped with an endoscopic grasper and placed under endoscopic view. Endoscopic placement took place via oral intubation of the esophagus with finally oro-nasal redirection and fixation with plasters.

OFD: The OFD for endoluminal therapy is handmade, as previously described, by wrapping a thin open-pore double-layered drainage film (Suprasorb® CNP, Drainage Film; Lohmann & Rauscher International GmbH & Co.KG, Rengsdorf, Germany) on the distal end of a small caliber redon drain, a gastric tube or the gastric segment of a naso-jejunal feeding tube (Freka® Trelumina, Fresenius Kabi Deutschland GmbH, Bad Homburg Germany). Sutures (MersileneTM, Polyester, 4 Ph. Eur., Ethicon®, Norderstedt, Germany) were used for the fixation of the drainage film around the tube. Drain insertion took place via nasal positioning and endoscopic guiding with grasper. Venting tubes in tri-lumen enteral feeding tubes has to be closed for ENPT.

Controlled Negative Pressure: A continuous vacuum of -125 mmHg is generated by electronic vacuum devices (KCI V.A.C. Ulta or V.A.C. Freedom; KCI USA Inc., San Antonio, TX, USA).

Procedural informations: In patients with suspected EJAL first an index endoscopy under general anesthesia with endotracheal intubation was indicated. Standard gastroscopes with outer diameter of 9.8mm were used with carbon dioxide insufflation.

Definition of a anastomotic leak were endoscopic or radiological dehiscences at the esophagojejunostomy with extravasation of fluids and gas.

Decision criteria for placement of OPD or OFD were the defect size, radiological findings and clinical situation of the patient. A CT scan in patients with suspected EJAL was done in all cases.

Re-endoscopy was performed after 3-7 days. In the case of persisting leak or in the case of uncertainty, the new ENPT system was re-inserted and treatment was continued. In patients with OPD change interval was 3-4 days, in patients treated with OFD interval was longer up to 7 days. Success was defined as complete closure of the perforation.

In patients with a good clinical situation with endoluminale placed OFD swallow of liquids is allowed.

Database:

An analysis was performed using SPSS v. 24.0.0.1 (IBM, Armonk, NY, USA). Data were presented as means ± SD.

Results Eight patients (4 females and 4 males with a mean age of 61.39 ± 12.92 years) were treated with ENPT for EJL. Patient's characteristics are presented in Table 2.

Mean time point of diagnosis the EJAL was day 6.25 ± 2.54 after resection. Three patients were treated at the ICU at the time of diagnosis of the EJAL. Symptoms that caused suspicion of EJAL were respiratory insufficiency, conspicuous secretion via drains, fever, and elevated inflammatory markers. All patients were treated and observed on ICU after detection an start of ENPT.

Findings of the index endoscopy varied strongly. Circumscribed insufficiencies, large leakages with secretion of putrid fluids or fibrin coated anastomosis with exposed clamps were seen. In Figure 1 and 2 examples of endoscopic finding during the index endoscopy are presented.

First treatment mode in all patients with EJAL was endoluminale ENPT. In five patients ENPT was performed with OPD and in three patients with OFD. In one obese patient with a complete anastomotic avulsion ENPT was changed to SEMS-therapy. Treatment characteristics are summarized in Table 3.

In order to achieve sepsis control additional surgery was indicated in seven of eight patients. Number of needed re-operations varied strongly.

Enteral feeding was established in all patients. Enteral feeding was ensured by nutrition tubes combined with ENPT through OFD in five patients and via needle catheter jejunostomy in three patients.

In seven patients treated with ENPT for EJAL therapy combined with surgery for sepsis control was successful. In five final endoscopic reports any dehiscences or insufficiencies were characterized and in two reports small and clean insufficiencies with good wound granulation were described.

A later endoscopic intervention of a post-treatment stenosis of the anastomosis was not detected in the analyzed patients.

Conclusion ENPT is a promising tool for treating EJAL. Furthermore, comparative studies between ENPT and other endoscopic treatment options for EJAL are needed to determine the best management options and indications for combined surgical interventions.

We recommend ENPT in endoluminal position in patients who suffered from EJAL combined with additional surgery if required to treat pleural or abdominal septic collections.

ELIGIBILITY:
Inclusion Criteria:

* anastomotic leak after oncological gastrectomy

Exclusion Criteria:

* all other patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
mortality rate | 30 days after surgery
  death by anastomotic leak

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No